CLINICAL TRIAL: NCT01572961
Title: Amélioration Des Techniques d'étude de la Micro-cirulation cutanée Chez Des Sujets Sains
Brief Title: Microvascular Function Assessment in Healthy Subjects
Acronym: MICROTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2010-10
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Physiology of Microvascular Skin
Keywords: Laser Doppler flowmetry, skin, microcirculation
MeSH Terms: interventions — Aspirin; acetylsalicylic acid lysinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Aspirin
  Interventions: Drug: acetylsalicilic acids (Aspirin)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acetylsalicilic acids (Aspirin) — single oral dose of 1g.
  Other Names: Aspegic 1000mg, sanofi aventis.
  Arms: Aspirin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Current stimulation induces microvascular dilation in human skin. The investigators aimed to study (1) whether the current vasodilation is amplified after two segmental current stimulation as compared to one stimulation; (2) whether this amplification relies on prostaglandin-sensitive mechanisms. A double-blind randomized placebo-controlled crossover trial is conducted in Angers, France.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years old
* Healthy subjects

Exclusion Criteria:

* Aspirin allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The increase of Laser Doppler Blood Flow after the second current stimulation | 1 hour

SECONDARY OUTCOMES:
The increase of Laser Doppler Blood Flow after the second current stimulation after aspirin administration | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mahe, M.D., Ph.D., Principal Investigator — University hospital of Angers
Locations (1):
- University Hospital, Angers, Maine et Loire, France

REFERENCES:
- [Derived] Mahe G, Abraham P, Humeau-Heurtier A, Gascoin L, Leftheriotis G, Durand S. Evidence for a vasomotor cyclo-oxygenase dependent mechanism of sensitization at the cutaneous level. Br J Clin Pharmacol. 2015 Aug;80(2):185-92. doi: 10.1111/bcp.12623. Epub 2015 May 26. PMID 25753207